CLINICAL TRIAL: NCT02136537
Title: Electrical Stimulation in Peripheral Arterial Disease
Acronym: PAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Member of staff moved on to training post. Trial halted and terminated
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/LO/0854; 14HH2054 (Other: Imperial College JRCO)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best medical therapy (Active Comparator): Claudicants treated according to local protocol - no added treatment
  Interventions: Other: Best medical therapy
- Best medical therapy plus NMES (Experimental): In addition to best medical therapy, subjects will receive bilateral neuromuscular stimulation of their legs, 4 hours per day.
  Interventions: Device: Bilateral NMES legs; Other: Best medical therapy

INTERVENTIONS:
Device: Bilateral NMES legs — Stimulation with the geko(TM) device, Firstkind Ltd, UK. 4 hours per day, bilateral, applied to the skin overlying the common peroneal nerve
  Arms: Best medical therapy plus NMES
Other: Best medical therapy — Treated according to local NHS protocol. At Imperial College Healthcare Trust, this will include diagnostic tests (medical interview and examination, ultrasound of blood vessels, diagnostic treadmill test, blood tests and Xrays as appropriate). This also includes lifestyle advice, treatment with appropriate drugs such as aspirin and statins, and supervised exercise.

SUMMARY:
The investigators wish to investigate the effects of neuromuscular stimulation on intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stable intermittent claudication (>6 months) with confirmation by medical imaging
* ABPI<0.9
* Absolute walking distance <500m

Exclusion Criteria:

* Pregnancy
* Cardiac pacemaker
* Previous lower limb major amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Absolute walking distance | 6 weeks
  Treadmill test (2mph, 0% grade increased by 3.5% every 3 minutes to a maximum of 15%

SECONDARY OUTCOMES:
Claudication distance | 6 weeks
  Treadmill test (as per absolute walking distance)

CONTACTS AND LOCATIONS:
Overall Officials: AH Davies, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom